CLINICAL TRIAL: NCT00298142
Title: A Prospective Randomised Clinical Trial to Investigate the Management of Headache Disorders. Study to Identify Prognostic Patient Characteristics and to Investigate the Additional Value of Physio-/Manual Therapy
Brief Title: Management of Headache Disorders: A Clinical Trial Screening for Prognostic Patient Characteristics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Hogeschool Antwerpen (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Headache Trial; OZR-VUB 997; OZR-HA G 815
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Headache
Keywords: Cervicogenic Headache; Migraine; Tension Type Headache
MeSH Terms: conditions — Headache; Post-Traumatic Headache; Migraine Disorders; Tension-Type Headache | interventions — Neurologists; Musculoskeletal Manipulations

INTERVENTIONS:
Procedure: Usual Care provided by a medical doctor (GP or Neurologist)
Procedure: Usual care plus Physio-/ Manual Therapy

SUMMARY:
The management of headache disorders is too often based upon trial and error or on personal beliefs and opinions. Seldom it is based on scientific arguments. Therefore the identification of prognostic patient characteristics is mandatory as this will lead to a more precise referral of headache patients.A prospective cohortstudy is designed to identify these prognostic patient characteristics. After testing, 186 headache patients (migraine, tension type headache and cervicogenic headache) will be randomly allocated to one of two treatment groups. Testing includes the fulfillment of questionnaires (Headache Diagnosis Questionnaire, Headache Inventory Questionnaire and the Headache Impact Test) and physical tests (Thermal Stimuli, Cervical Spine examination and Pressure Algometry). Treatment groups are a usual care group (administered by a medical doctor) and a usual care plus physio-/ manual therapy treatment. After six weeks of treatment subjects will complete the headache inventory list and the Headache Impact Test a second time. The perceived effect will be registered allowing the distinction between responders (positive effect) and non-responders (no effect or worse). Logistic regression-analysis will be used to identify the specific patient characteristics of the responders and the non-responders. Secondly the additional value of the physio-/ manual therapy intervention will be examined. Follow-up measurements up to 52 weeks are provided.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking
* Willing to participate
* At least 18 years old
* Combination of headache and neck pain
* Headache since at least two months and at least twice a month
* A combination of migraine, tension type headache and cervicogenic headache

Exclusion Criteria:

* Clusterheadache
* Trigeminusneuralgia
* Peripheral neuropathy
* A history with neck surgery
* Comorbidity with chronic muskuloskeletal pain like fibromyalgia
* Radicular pain in the upper extremity
* Osteoarthritis
* Down Syndroom
* Physio/ manual therapy treatment in the last 12 months for this headache complaint.
* The use of prescribed medication (like NSAIDs and triptans) for this headache complaint during the last two months
* Pregnancy
* Red flags as described in the Dutch General Practitioners Headache Guideline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Manual Examination of the Cervical Spine
Pressure algometry
Thermal stimulation
Perceived effect
HIT-6

SECONDARY OUTCOMES:
Frequency of headache
Intensity of headache
Medication Intake
Additional Profession help
Absenteism

CONTACTS AND LOCATIONS:
Overall Officials: Willem De Hertogh, MSc, Principal Investigator — Vrije Universiteit Brussel
Locations (14):
- Belgium (14):
  - UZA - Neurology Dept., Antwerp, Antwerp
  - AZ-VUB, Brussels, Brussels Capital
  - GP-De Loof, Aalst
  - GP-Roelants, Boom
  - GP-Marmitte, Dilbeek
  - GP - Sengeleng, Hamme
  - GP-De Hertogh, Kampenhout
  - GP- De Smet, De Leu, Van Watermeulen, Thienpont, Wille, Laarne
  - GP - Riffi Abdellatif, Mechelen
  - GP-Vande Voorde, Merchtem
  - GP - Goossens, Reet
  - GP- Dingemans, Michiels, Declercq, Reet
  - GP-Van de Heijning, Schoten
  - GP-Roelands, Zemst

REFERENCES:
- [Background] De Hertogh WJ, Vaes PH, Vijverman V, De Cordt A, Duquet W. The clinical examination of neck pain patients: the validity of a group of tests. Man Ther. 2007 Feb;12(1):50-5. doi: 10.1016/j.math.2006.02.007. PMID 16769236
- [Background] De Hertogh WJ, Vaes PH, Devroey D, Truijen S, Duquet W, Oostendorp R. Management of headache disorders: design of a randomised clinical trial screening for prognostic patient characteristics. BMC Musculoskelet Disord. 2007 Apr 26;8:38. doi: 10.1186/1471-2474-8-38. PMID 17462091
- [Result] De Hertogh W, Vaes P, Devroey D, Louis P, Carpay H, Truijen S, Duquet W, Oostendorp R. Preliminary results, methodological considerations and recruitment difficulties of a randomised clinical trial comparing two treatment regimens for patients with headache and neck pain. BMC Musculoskelet Disord. 2009 Sep 23;10:115. doi: 10.1186/1471-2474-10-115. PMID 19775434